CLINICAL TRIAL: NCT06400056
Title: Clinical and Laboratory Evaluation of Antifungal Resistance in Tinea Capitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Atef Ibrahim, Dermatologist, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Fungal resistance
Record Dates: First submitted 2023-03-18; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Fungal Resistance
MeSH Terms: interventions — Terbinafine

STUDY DESIGN:
Intervention Model Description: More than 4 years old
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Terbinafine (Experimental): Patients will be treated by systemic terbinafine alone for 6 weeks
  • Dosage: 25 kg for 125 mg 25-35 kg for 187.5 mg 35 for 250 mg
  Interventions: Drug: Terbinafine

INTERVENTIONS:
Drug: Terbinafine — FDA approved

SUMMARY:
AIM OF WORK :

1. Detect the most common fungal strains that cause tinea capitis
2. Detect Different effectiveness of terbinafine in different cases
3. Detect the resistant strains.
4. Detect the mycological and the clinical cure rates upon using systemic terbinafine in treatment of tinea capitis

DETAILED DESCRIPTION:
Introduction:

* Tinea capitis is a superficial fungal infection of the skin of the scalp, with a propensity for attacking hair shafts and follicles . The disease is considered to be a form of superficial mycosis or dermatophytosis
* It may affect all or part of the child's scalp.
* Mold-like fungi called dermatophytes cause tinea capitis ,It is caused primarily by Dermatophyte species Microsporm and trichopyton,, In Egypt, dermatophytes called Microsporum canis and Microsporum audouinii are the most common causes of the infection. Fungi thrive in warm, moist environments. It commonly grows in tropical places.
* Tinea capitis can be divided into inflammatory and non-inflammatory types, the non-inflammatory type usuallywill not be complicated by scaring alopecia , the inflammatory type may result in Kerion ,a painful nodule with pus and scaring alopecia, The clinical manifestations of tinea capitis are classified as endothrix, ectothrix, or favus. In the endothrix form, hyphae grow down the follicle and penetrate the hair shaft, then grow completely within the hair shaft. This form is caused predominantly by T. tonsurans and T. violaceum In the ectothrix form, the hyphae invade the hair shaft at mid follicle. Afterwards, hyphae grow out of the follicle covering the hair surface. This form is caused by M. canis, M. audouinii, Microsporum ferrugineum, and Trichophyton verrucosum. The hyphae grow parallel to the hair shaft in favus form then degenerate, leaving long tunnels within the hair shaft. Favus form is caused by Trichophyton schoenleinii and is characterized by yellow crust around the hair shafts and can result in permanent scarring alopecia.
* ♦ Tinea capitis also spreads very easily. The patients can catch the infection from contact with infected people, animals and soil. They can also get it by using objects and touching surfaces that harbor the fungus. Tinea capitis can live for a long time on infected objects and surfaces. It is very contagious and can spread quickly among children
* The diagnosis is suspected primarily clinically based on the appearance of the scalp lesion. A Wood's lamp test performed to confirm the presence of a fungal scalp infection , Dermoscopy is a useful and non invasive diagnostic tool which aids in the diagnosis of tinea capitis ,the diagnosis can be confirmed by microscopic examination of KOH,
* Fungal culture is the gold standard to diagnose dermatophytosis,
* fungal culture can help to differentiate fungal species
* The treatment of tinea capitis requires systemic antifungal therapy because topical antifungal agents cannot penetrate the hair shaft sufficiently to eradicate infection. Griseofulvin, the former gold standard agent, has been associated with treatment failure; a retrospective review of patients' medical records revealed a failure rate of 39.3% , in octobr 2007 The FDA has approved terbinafine oral granules (Lamisil), which can be sprinkled on food, for tinia capitis in children four years and older , fluconazole and Itraconazole also used in treatment of Tinea capitis although they are not FDA approved
* In the past few years , Numerous cases of tinea capitis that was initially resistant to systemic antifungal or recurred rapidly after a brief interval improvement recently have been seen
* In general, clinical resistance is considered to be the persistence or progression of an infection despite appropriate antimicrobial therapy , This resistance can be attributed to a combination of factors related to the host, the antifungal agent, or the pathogen .

ELIGIBILITY:
Inclusion Criteria:

* patients from both sexes aged > 4 years old.
* patients have tinea capitis (scaly type)

Exclusion Criteria:

* Patients have other types of tinea capitis infection.
* Patients with heart valve diseases , Hearing loss , liver or kidney diseases.
* Pregnant or lactating females.
* Personal or family history of malignancy.
* Immunocompramised patients.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
-Detect the most common Fungal strains that cause tinea capitis | Baseline
  * Detect the most common Fungal strains that cause tinea capitis by doing :
  * Fungal culture after gentle scraping of surface of affected area.
Resistant strain in tinea capitis | Baseline
  - Detect the resistant strain by using culture of scrapped sample.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Moubasher, Professor, Study Director — Supervisor; Radwa Bakr, Professor, Study Director — Supervisor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelt L, Nenoff P, Uhrlass S, Kruger C, Kuhn P, Eichhorn K, Buder S, Beissert S, Abraham S, Aschoff R, Bauer A. [Terbinafine-resistant dermatophytoses and onychomycosis due to Trichophyton rubrum]. Hautarzt. 2021 Oct;72(10):868-877. doi: 10.1007/s00105-021-04879-1. Epub 2021 Aug 30. German. PMID 34459941
- [Background] Hawks MK, Rupert JP, Svarverud JE. Terbinafine for Onychomycosis. Am Fam Physician. 2018 Aug 1;98(3):Online. No abstract available. PMID 30215902
- [Background] Lian LD, Shi LY, Zhu J, Liu R, Shi L, Ren A, Yu HS, Zhao MW. GlSwi6 Positively Regulates Cellulase and Xylanase Activities through Intracellular Ca2+ Signaling in Ganoderma lucidum. J Fungi (Basel). 2022 Feb 14;8(2):187. doi: 10.3390/jof8020187. PMID 35205940
- [Result] Moreno-Sabater A, Normand AC, Bidaud AL, Cremer G, Foulet F, Brun S, Bonnal C, Ait-Ammar N, Jabet A, Ayachi A, Piarroux R, Botterel F, Houze S, Desoubeaux G, Hennequin C, Dannaoui E. Terbinafine Resistance in Dermatophytes: A French Multicenter Prospective Study. J Fungi (Basel). 2022 Feb 23;8(3):220. doi: 10.3390/jof8030220. PMID 35330222